CLINICAL TRIAL: NCT05936918
Title: Effects of Transcutaneous Electrical Acupoint Stimulation Combined With Transverse Abdominis Plane Block on Perioperative Pain and Early Postoperative Recovery in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Application of Transcutaneous Electrical Acupoint Stimulation in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Wang wanxia, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-YKL04- (ke04)
Record Dates: First submitted 2023-06-06; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Pain Postoperative; Postoperative Recovery
Keywords: Transcutaneous electrical acupoint stimulation; Postoperative pain; Visceral pain; Early recovery after surgery
MeSH Terms: conditions — Pain, Postoperative; Visceral Pain

STUDY DESIGN:
Intervention Model Description: The study was primarily a randomized controlled study in which patients were randomly assigned to each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data collector
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TT group (Experimental): Bilateral Neiguan acupuncture points (PC6), Hegu acupuncture points (LI4), Zusanli (ST36) were selected, and percutaneous acupuncture points were electrically stimulated with electronic acupuncture equipment 30min before anesthesia, and then bilateral abdominal transverse plane blockade was performed
  Interventions: Other: Transcutaneous electrical acupoint stimulatios; Other: Bilateral transverse abdominal plane block
- TE group (Active Comparator): Bilateral Neiguan acupuncture points (PC6), Hegu acupuncture points (LI4), Zusanli (ST36) were selected, and percutaneous acupuncture points were electrically stimulated with electronic acupuncture equipment 30min before anesthesia
  Interventions: Other: Transcutaneous electrical acupoint stimulatios
- TA group (Active Comparator): Bilateral transverse abdominal plane block is performed prior to anesthesia
  Interventions: Other: Bilateral transverse abdominal plane block
- C group (No Intervention): Percutaneous electrical stimulation of acupoints and transverse abdominis plane block are not permitted before anesthesia

INTERVENTIONS:
Other: Transcutaneous electrical acupoint stimulatios — Percutaneous electrical stimulation technology of acupuncture points is a technology that uses a trace current close to human bioelectricity on the surface of acupuncture points to prevent and treat diseases guided by meridian theory, and is a new treatment of percutaneous nerve electrical stimulation combined with acupuncture points. As one of the related techniques of acupuncture, it is a safe, non-invasive, simple and new acupoint stimulation method
  Arms: TE group; TT group
Other: Bilateral transverse abdominal plane block — Transverse abdominis plane block is a technique in which a local anesthetic is injected into the transverse abdominis plane to block sensory nerves passing through this plane to achieve analgesic effect
  Arms: TA group; TT group

SUMMARY:
To explore the application of transcutaneous electrical acupoint stimulation combined with transverse abdominis plane block in Laparoscopic cholecystectomy, in order to reduce postoperative pain and promote postoperative recovery.

DETAILED DESCRIPTION:
Percutaneous electrical acupoint stimulation has been applied in preoperative prophylaxis, intraoperative anesthesia and postoperative rehabilitation, and can reduce perioperative anxiety, improve the efficacy of preoperative smoking cessation and alcohol abstinence, and shorten the preoperative fasting time. During surgery, it can reduce the amount of anesthetic drugs, anti-inflammatory and anti-stress effects, stabilize circulation, and protect important organs; After surgery, improve the speed and quality of wake-up of patients, promote the recovery of maintenance function, regulate immune function, and reduce postoperative adverse reactions such as postoperative pain, postoperative nausea and vomiting, postoperative urinary retention, etc. As one of the common nerve blocks, transverse abdominis block is used clinically, and its main function is to relieve perioperative pain and reduce the amount of traumatic stress and analgesic drugs

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I and II
* Age 18-65 years
* Laparoscopic cholecystectomy for the first time
* There is no rupture, infection in the acupoint pasting site
* The patient knows and signs the informed consent form

Exclusion Criteria:

* People with visual impairment, hearing impairment and alcoholism
* History of diabetes, myocardial infarction or cerebrovascular accident, liver and kidney dysfunction
* Those who are allergic to non-steroidal drugs, anticholinergic drugs, and anesthetic drugs
* Those who are unable to cooperate or refuse to participate in the research or request to withdraw during the research process
* Those with contraindications to percutaneous electrical stimulation, including local skin damage, infection or implantation of electrophysiological devices in the body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-02 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS(visual analogue scale) score | The day before surgery
  Postoperative pain is assessed after surgery by using visual analogue scoring. A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.
VAS(visual analogue scale) score | After the operation 30minute
  Postoperative pain is assessed after surgery by using visual analogue scoring. A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.
VAS(visual analogue scale) score | After the operation 6hour
  Postoperative pain is assessed after surgery by using visual analogue scoring. A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.
VAS(visual analogue scale) score | After the operation 12hour
  Postoperative pain is assessed after surgery by using visual analogue scoring. A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.
VAS(visual analogue scale) score | After the operation 24hour
  Postoperative pain is assessed after surgery by using visual analogue scoring. A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.
VAS(visual analogue scale) score | After the operation 48hour
  Postoperative pain is assessed after surgery by using visual analogue scoring. A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | The day before surgery; After the operation 24hours, 48hours
  After surgery, patients are asked about nausea and vomiting. Postoperative nausea and vomiting is assessed after surgery by using visual analogue scoring. Using a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no nausea and vomiting, and 10 points represent the most severe nausea and vomiting that is unbearable.
Early postoperative recovery of quality | The day before surgery; After the operation 24hours, 48hours
  The quality of early postoperative recovery was assessed using The Quality of Recovery-15 scale after surgery, scores range from 0 (QoR very poor) to 150 (QoR excellent), with higher scores representing better quality of recovery
Exhaust and bowel movements | After the operation 24hours, 48hours
  Record the time of the patient's first exhaust bowel movement after surgery
Concentration of serum interleukin-6 | the day before surgery; When entering the operating room; 10minutes after peeling; 5 minutes after the operation; The first day after surgery
  Perioperative venous blood was drawn to detect serum interleukin-6
Concentration of serum cortisol | the day before surgery; When entering the operating room; 10minutes after peeling; 5 minutes after the operation; The first day after surgery
  Perioperative venous blood was drawn to detect serum cortisol
Concentration of serum C-reactive protein | the day before surgery; When entering the operating room; 10minutes after peeling; 5 minutes after the operation; The first day after surgery
  Perioperative venous blood was drawn to detect serum C-reactive protein